CLINICAL TRIAL: NCT00163072
Title: Pharmacokinetics and Safety of Transdermal Megestrol Acetate
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Andrew S. Freiberg, MD, Penn State University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM IRB# 18400
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2007-04

CONDITIONS: Cachexia
Keywords: transdermal; Megace; pharmacokinetics
MeSH Terms: conditions — Cachexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: transdermal Megace — oral vs transdermal levels

SUMMARY:
Rationale: Megestrol acetate (Megace®) is a progestin analog that is FDA approved for the palliative treatment of breast and endometrial carcinoma. It is also commonly used as an appetite stimulant, particularly in HIV and cancer patients with poor appetite from their primary disease and/or their therapy. Megace is well absorbed orally, however, many patients, particularly younger ones have difficulty taking oral medications. Transdermal progestins are available and are FDA approved. For example, Ortho EvraTM is a transdermal contraceptive patch containing an estrogen (ethinyl estradiol) and a progestin (norelgestromin).

Key Objectives: Compare the pharmacokinetics of orally administered vs. transdermal Megace and determine if there are any local side effects of the transdermal route.

DETAILED DESCRIPTION:
Study Population: Patients of any age who are already receiving oral Megace as an appetite stimulant. Patients must have an indwelling IV catheter in order to draw drug levels.

Major Inclusion & Exclusion Criteria: Known hypersensitivity to the transdermal vehicle. Taking any other medicine that would interfere with the Megace assay. Weight less than 10 kg.

Allocation to Groups: Patients will serve as their own controls.

Summary of Procedures: Patients will be on a stable dose of oral Megace. To determine the steady state peak level and half-life for each patient, blood (2cc) will be drawn for a level in clinic 3 hours after an oral dose, then daily for 1-3 days. Patients may then resume their oral Megace, but must stop the medicine at least 5 half-lives prior to the transdermal dose. The transdermal dose will be applied as a gel under a transparent patch in clinic, and blood will be collected prior to, 10, 30, 60, 90, and 120 minutes, and 4 hours after the dose. The patch will be removed after the 4 hour blood level. The patient will return the following day for a 24 hour level, and the patient will be examined briefly for any local effects of the drug or vehicle, and then may resume the oral dose.

Major Risks & Discomforts: Patients will need to be in clinic for 3-5 separate days, one of which will last at least 4 hours, for drug levels to be drawn. There may be mild skin reaction to the transdermal vehicle or the Megace.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any age who are already receiving oral Megace as an appetite stimulant.
* Patients must have an indwelling IV catheter in order to draw drug levels.

Exclusion Criteria:

* Known hypersensitivity to the transdermal vehicle.
* Taking any other medicine that would interfere with the Megace assay.
* Weight less than 10 kg.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-10; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
pharmacokinetics | 2 months
safety | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S Freiberg, MD, Principal Investigator — Penn State University
Locations (1):
- Hershey Medical Center, Hershey, Pennsylvania, United States